CLINICAL TRIAL: NCT04558086
Title: The Effects of Using an Interactive Game With Virtual Reality to Reduce the Pain and Fear for Children During an Intravenous Placement
Brief Title: The Effects of Using an Interactive Game With Virtual Reality for Children During Intravenous Placement
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: National Yang Ming Chiao Tung University (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Supportive Care
Other Study IDs: 108163-F
Record Dates: First submitted 2020-09-16; First posted 2020-09-22 (Actual); Last update posted 2020-09-22 (Actual); Status verified 2020-09

CONDITIONS: Pian; Fear
Keywords: Therapeutic play,virtual reality, intravenous placement, school-age, pain, fear
MeSH Terms: conditions — Yaws; Pain

STUDY DESIGN:
Who Masked: Participant
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Reduce pain and fear (Experimental): To develop the intervention strategies of hospitalized school-age children with IV placement, using interactive virtual reality(VR)as a guiding play and emotional catharsis play, to further examine the effectiveness of reducing IV pain and fear.
  Interventions: Device: Virtual reality
- control group (Experimental): To develop the intervention strategies of hospitalized school-age children with IV placement, using photo book to further examine the effectiveness of reducing IV pain and fear.
  Interventions: Device: Photo book

INTERVENTIONS:
Device: Virtual reality — To develop the intervention strategies of hospitalized school-age children with IV placement, using interactive virtual reality(VR)as a guiding play and emotional catharsis play, to further examine the effectiveness of reducing IV pain and fear.
  Arms: Reduce pain and fear
Device: Photo book — To develop the intervention strategies of hospitalized school-age children with IV placement, using Photo book to further examine the effectiveness of reducing IV pain and fear.
  Arms: control group

SUMMARY:
To develop the intervention strategies of hospitalized school-age children with IV placement, using interactive virtual reality(VR)as a guiding play and emotional catharsis play, to further examine the effectiveness of reducing IV pain and fear.

ELIGIBILITY:
Inclusion Criteria:

* Children ages 6-12.
* Children who where clearly conscious.
* Children who agreed and were required to receive intravenous injections after physicians' diagnoses.
* Children and their primary caregivers who could communicate in Mandarin or Taiwanese
* Children and their primary caregivers who could read Chinese that agreed to participate in this study and sign written consent forms

Exclusion Criteria:

* Children with developmental delay, epilepsy, or heart diseases
* Children undergoing chemotherapy; children who were visually or hearing impaired
* Children who were nearsighted with more than 8.0 diopters or farsighted with 5.0 diopters.
* Children who had sustained head trauma in the past month
* Children who were confirmed to be obese according to the recommended body mass index values for children and adolescents
* Children who required blood transfusions and blood preparation to be performed according to physician diagnoses
* Children who received two or more intravenous injections and had their blood drawn only one time

Ages: 6 Years to 12 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child
Enrollment: 134 (Actual)
Dates: Start 2020-06-05 (Actual); Primary Completion 2020-09-11 (Actual); Study Completion 2020-09-11 (Actual)

PRIMARY OUTCOMES:
The degrees of pain experienced by the children. | The posttests 8 min after the tourniquets were worn.
  Measurement of pin using the Wong-Baker Faces Pain Rating Scale (WBFPS). The scale contains six cartoon faces shwing pain ratings of 0~10, which are, from left to right, no pain(0), a little pain (2), mild pain (4), average pain (6), severe pain (8), and excruciating pain (10).The children, primary caregivers, and nurses were asked to select the faces that best described the pain levels experienced by the children receiving intravenous injections; the pain levels were subsequently converted into numerical values .
The degrees of fear experienced by the children. | The posttests 8 min after the tourniquets were worn.
  Measurement of fear using the Choldren Fear Scale(CFS).The scale consists of five cartoon faces showing fear ratings of 0-4, which were no fear (0), a little fear (1), some fear (2), very fear(3) and extreme fear (4). The children, primary caregivers, and nurses were asked to select the faces that best described the fear levels of the children receiving intravenous injections. The pain levels were subsequently converted into numerical values.

CONTACTS AND LOCATIONS:
Locations (1):
- National Yang-Ming University, Taipei County, Taiwan